CLINICAL TRIAL: NCT04103047
Title: Temporomandibular Joint (TMJ) Dysfunction Following the Use of Supraglottic Airway Devices
Brief Title: TMJ Dysfunction Following Use of SAD
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 262069
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Temporomandibular Joint Disorder Bilateral
Keywords: Temporomandibular joint disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SAD group: Adult surgical patients who are due to undergo general anaesthesia and requiring SAD insertion will be identified on the day of surgery.
  Interventions: Other: SAD

INTERVENTIONS:
Other: SAD — The patients who have an SAD inserted as part of their normal Anaesthetic plan will be consented prior to their Anaesthetic and then have a questionnaire to fill out post operatively.

SUMMARY:
The aim of this study is to assess how the use of a breathing tube (Supraglottic Airway Device) can affect the function of the jaw joint (Temporomandibular joint) movement. This type of breathing tube is used for nearly 60% of general anaesthetics. To facilitate insertion of this breathing tube, assisted mouth opening and forward movement of the jaw are required.

These movements occur at the jaw joint (temporomandibular joint). In addition, for the duration of the operation the mouth is kept slightly open by a breathing tube. There are a few case reports in the literature suggesting minor effect on the jaw joint. Therefore, we wish to study this further by evaluating the function of the jaw joint, 4 to 24 hours after the operation.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1 Background Supraglottic airway devices (SADs) are part of the mainstay of anaesthetic practice, being the primary airway management device in 56% of general anaesthetics. SADs are used by both novice and experienced anaesthetists, in addition to anaesthetic practitioners, non-anaesthetic clinicians and other health care professionals. They are routinely used to deliver anaesthetic gases and oxygen to the patient during general anaesthesia. In an airway emergency, for example in the case of failed intubation, a second-generation SAD has been recommended as a rescue device to maintain oxygenation. This can also then be used as a conduit to intubate the trachea.

   Although insertion of SADs considered to be relatively easy, it requires certain manoeuvres. These include extension of the head and neck flexion, use of a jaw thrust with adequate mouth opening, and then introduction of the device with a firm and gentle motion down and backwards along the hard palate. These methods are thought to improve the time to successful insertion of the SAD. Whilst movements such as these can be viewed as simple and 'benign', investigators are concerned that these can cause dysfunction of temporomandibular joint dysfunction in the postoperative period.

   Most published research has been focused on insertion success and time taken to insert the device. There has been limited research and literature about complications following SAD insertion, such as gastric aspiration, trauma to or loss of the airway, and about best insertion techniques, as mentioned above, including use of thermally softened SADs.

   However, there are few reports of TMJ dysfunction and dislocation following SAD insertion under general anaesthesia. This may be due in part to general anaesthesia causing reduced muscle tone and greater joint mobility, but investigators assume a degree of dysfunction is due to passive manipulation of the TMJ with forward movement of the jaw and widened mouth opening for a prolonged period of time.

   Some TMJ dysfunction may also be attributed to use of the SAD itself being in situ for a prolonged period, where the cuff of the device occupies the oropharynx causing forward displacement of the jaw. The recommended duration of SAD insertion ranges from one to four hours.

   1.2 Proposed study This study aims to evaluate the degree of TMJ dysfunction in the postoperative period, in patients where a SAD has been used a primary airway device. The study will be conducted at University Hospitals Coventry and Warwickshire National Health Service (NHS) Trust and Birmingham Heartlands Hospital, part of the University Hospital of Birmingham NHS Trust.

   A member of the research team will approach eligible patients preoperatively to explain the study, provide written information and obtain written consent. Consenting participants will then be asked to complete a questionnaire and the member of the research team will measure and record an airway assessment including jaw movements. Post anaesthesia, participants will again be approached to complete a questionnaire and the research team member will re-measure jaw movements. The preoperative responses and measurements will be compared with those of postoperative responses and measurements.

   1.3 Study population Those patients who undergo general anaesthesia for surgery, in whom the SAD will be used as the primary airway device.

   1.4 Treatment / Intervention (if applicable) The decision regarding the method of airway management is decided by the patient's responsible anaesthetist, according to the clinical indication. There is no additional treatment or intervention as a result of this study, it is purely observational.
2. RATIONALE 2.1 Aims and hypothesis The aim of this study is to assess for an objective difference between pre- and post-operative jaw movements following the use of SADs, and to identify any subjective discomfort or perceived difference in TMJ function.

2.2 Justification

SADs are commonly used in anaesthetic and non-anaesthetic practice. SADs are placed by clinicians of varying expertise, frequently using simple airway manoeuvres or the triple airway manoeuvre to aid correct placement. Historically research has been carried out regarding methods to aid correct SAD positioning and time to correct positioning, and also regarding complications following the use of SADs as reported in 4th national audit project of the Royal College of Anaesthetists and Difficult Airway Society. In recent years case reports have been published concerning TMJ dislocation and dysfunction after the use of the SAD.

are unaware of any studies investigating TMJ function after routine use of SAD under general anaesthesia. If there is a significant deterioration in the function of TMJ during postoperative period further guidance need to be devised on safe use of SADs. If there are no differences, this will reassure the common and routine practice of use of SADs. If a difference is found, it could lead to a change in education and improved clinical practice, ultimately enhancing patient safety.

2.3 Assessment and management of risk This study is of patients' pre- and post-operative TMJ function. Investigators will be approaching the patients in these periods to take part in completing a short questionnaire, and also taking measurements of jaw movements. Patient management will not be affected by the study. Investigators do not anticipate any additional risks or benefits to the patient.

4. STUDY DESIGN This is a semi-qualitative questionnaire study of patients to assess TMJ function after the airway has been secured with a SAD during general anaesthesia. The study protocol will be discussed with the local research and development department and appropriate Research Ethics Committee (REC) approval will be obtained.

Adult surgical patients who are due to undergo general anaesthesia and requiring SAD insertion will be identified on the day of surgery. These patients will then be approached and given patient information sheet. They will be given adequate time to read the information sheet and any questions will be answered.

Consenting patients will be asked to complete a pre-operative questionnaire and jaw movements (mouth opening = inter-incisor distance, jaw protrusion= the distance between the upper and lower incisors when the lower jaw is fully protruded) and lateral jaw movements = right and left lateral sliding of lower jaw = distance between upper and lower molars) will be measured by one of the research team member. The above procedure will be repeated 4 to 24 hours in the post-operative period using post-operative patient questionnaire and measurements of jaw movements.

Sample size From our previous research on evaluating the correlation between airway assessment parameters and depth of cricothyroid membrane, the observed mean for inter-incisor distance (IID) was 45.5 mm with standard deviation 8.1. Investigators considered a reduction in IID following used of SAD is clinically significant. Assuming a mean baseline IID of 35- 45 mm, with a pow-er of 90% power to detect a 10% reduction in IID with p<0.05, in total 120 patients were needed. Using G*Power 3.1.9.4 confirmed that a sample size of 120 using a paired t-test with 2 tails will allow detection of significant. In total, 130 patients will be recruited to overcome dropouts and incomplete data. Once screened, eligible patients will be given information leaflets explaining the reason for the study, and any questions answered. Following written consent, patients will be given a questionnaire to be completed and jaw movements as described above will be measured.

7. TRIAL PROCEDURES The suitable patients for the study will be screened from the operating theatre list. During the preoperative assessment one of the investigator or co-investigator will provide patient information sheet. Patients will be given adequate time to read the information and any questions will be answered. If they are satisfied and willing to take part in the study, written consent will be obtained.

7.1 Recruitment Both Chief investigator and co-investigators identify the suitable operating list. Then the suitable patients will be identified based on the scheduled surgical procedure. Only those patients meeting the inclusion criteria will be approached.

7.1.1 Patient identification

The patients undergoing surgery that requires tracheal intubation are suitable to be included in the study. Based on the scheduled surgery on the operating list, the suitable patients will be identified. During the preoperative assessment one of the investigator or co-investigator will provide patient information sheet. Patients will be given adequate time to read the information and any questions will be answered. If they are satisfied and willing to take part in the study, written consent will be obtained.

7.1.2 Payment There are no associated payments for participation in this study as no extra expenses are expected to be incurred by the participants.

7.2 Consent Participants will be given enough time to read the patient information leaflet (minimum of 2 hours). Once they have read the information, any questions will be answered. If they agree for the study, they will be asked to complete the consent form. The consent will be obtained by chief investigator, coinvestigator or one of the research team member, supervised by one of the investigator.

7.3 Baseline data Base line data includes gender, age, weight, height, BMI & American Society Anesthesiologist (ASA) score Airway assessment includes Mallampati score, thyromental distance, mouth opening and neck movement

7.4 Trial assessments Visit one - prior to anaesthesia

Using the patient questionnaire, the following will be recorded:

* Patient mouth opening and pain at the temporomandibular joint
* Yes and no answers to questions regarding TMJ function

A member of the research team will then record:

* Mouth opening = inter-incisor distance
* Jaw protrusion= the distance between the upper and lower incisors when the lower jaw is fully protruded
* Lateral jaw movements = right and left lateral sliding of lower jaw = distance between upper and lower molars on lateral sliding

Visit two: 4-24 hours post operatively

Using the patient questionnaire, the following will be recorded:

* Patient mouth opening and pain at the temporomandibular joint
* Yes and no answers to questions regarding TMJ function

A member of the research team will then record:

* Mouth opening = inter-incisor distance
* Jaw protrusion= the distance between the upper and lower incisors when the lower jaw is fully protruded
* Lateral jaw movements = right and left lateral sliding of lower jaw = distance between upper and lower molars on lateral sliding

7.5 Long term follow-up assessments There is no long term follow-up for this study. The participant will only be approached twice as described as above. Once pre-operatively and once postoperatively.

8. STATISTICS

8.1 Sample size calculation From our previous research on evaluating the correlation between airway assessment parameters and depth of cricothyroid membrane, the observed mean for inter-incisor distance (IID) was 45.5 mm with standard deviation 8.1. A 10% reduction in IID following use of SAD was considered to be clinically significant. Assuming a mean baseline IID of 35- 45 mm, with a power of 90% power to detect a 10% reduction in IID with p<0.05, a total of 120 patients are needed. Using G*Power 3.1.9.4 confirmed that a sample size of 120 using a paired t-test with 2 tails will allow detection of significant. Investigators aim to recruit 130 patients to overcome drop outs and incomplete data. Once screened, eligible patients will be given information leaflets explaining the reason for the study, and any questions answered. Following written consent, patients will be given a questionnaire to be completed and jaw movements as described above will be measured.

8.4 Participant population

All patients who are included in the study will be included in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* • All patients aged above 18, presenting for elective surgical procedure under general anaesthesia, where a supraglottic airway device can be used as primary airway device. This involves a group of patients presenting for day case surgical procedures.

Exclusion Criteria:

* • Patients under the age of 18

  * Patients who do not consent to being part of the study
  * Patients in whom SAD is unlikely to be the primary airway device
  * If a translator is not available at the time, participants who cannot reasonably read and communicate in English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 130 patients undergoing any operation where the Anaesthetist feels the best choice of airway management device is a supraglottic airway device.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Difference between preoperative and postoperative interincisor distance in mm | within 24 hours
  The primary outcome measure is the difference between preoperative and postoperative interincisor distance in mm. When mouth is fully opened, the distance between the incisor teeth is measured in mm. This measurement is repeated in the postoperative period between 4 to 24 hours after the surgery. The measurements will be done using TheraBite ruler (ATOS medical, Nottingham, UK). The data are compared using paired t test or Mann-Whitney U test.
Difference between preoperative and postoperative lateral jaw movement in mm | within 24 hours
  The difference between preoperative and postoperative lateral jaw movement in mm. Lateral movement of the lower jaw (the lateral sliding of midpoint of lower jaw in reference to midline is measured in mm. This reference is repeated in the postoperative period between 4 to 24 hours after the surgery. The measurements will be done using TheraBite ruler (ATOS medical, Nottingham, UK). The data are compared using paired t test or Mann-Whitney U test.

SECONDARY OUTCOMES:
Patient reported pain in the jaw joint (temporomandibular joint) | Within 24 hours
  Secondary outcomes will be the patient reported pain in the jaw joint (temporomandibular joint). During the preoperative period patient is asked to press on the jaw joint using index finger and record the pain experienced on visual analogue scale of 0 to10. The same is repeated in the postoperative period between 4 to 24 hours. Pain score will be compared using Mann-Whitney U test. The lower values represent better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
We aim to share the study protocol, the statistical analysis plan, informed consent form and study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of completion of recruitment of patients.
Access Criteria: We aim to publish our findings in an Anaesthetic journal.

REFERENCES:
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Michalek P, Donaldson W, Vobrubova E, Hakl M. Complications Associated with the Use of Supraglottic Airway Devices in Perioperative Medicine. Biomed Res Int. 2015;2015:746560. doi: 10.1155/2015/746560. Epub 2015 Dec 13. PMID 26783527
- [Background] Sia SL, Chang YL, Lee TM, Lai YY. Temporomandibular joint dislocation after laryngeal mask airway insertion. Acta Anaesthesiol Taiwan. 2008 Jun;46(2):82-5. doi: 10.1016/S1875-4597(08)60032-6. PMID 18593655
- See also: Using the i-gel® supraglottic airway - Intersurgical — https://www.intersurgical.com/content/files/61747/-1200643841
- See also: TMJ scale — https://www.tmjscale.com/pdf_docs/TMJForm.pdf